CLINICAL TRIAL: NCT04511780
Title: Psychological Impact of COVID-19 Outbreak on Caregivers Involved in Intensive Care Unit Patient Management: Impact on the Occurrence of Post-traumatic Stress Disorder, Anxiety, Depression and Burn Out Syndrome
Brief Title: Psychological Impact of COVID-19 Outbreak on Caregivers
Acronym: PSY-CO-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2020/JYL-03
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Covid19; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Critical Illness; COVID-19; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: • Caregivers (doctors senior and junior, nurses, aid nurses) involved in the staff (permanent or transient, full or partial time) of ICU patients during Covid-19 outbreak
  Interventions: Other: questionnaire filling

INTERVENTIONS:
Other: questionnaire filling — assessment of post-traumatic stress, anxiety and burn out

SUMMARY:
Based on the experience of previous pandemics, countries reacted by applying different upgrade strategies to prevent or delay the widespread of the disease. Therefore, measures such as border closure, school closure, restrict social gathering (even shutdown of workplaces), limit population movements, and confinement meaning quarantines at the scale of cities or regions. In public hospitals, several measures have been decided to concentrate the power of care on potential wave of admissions of patients with severe forms of Covid-19. In this purpose, the number of available beds in Intensive Care Units (ICU) has been increased by two-fold and scheduled non-emergency surgical procedure have been cancelled. That means:

1. For the most severe patients, new personals (physician such as anesthesiologists, nurses of other units) have been transferred in ICUs.
2. For the less severe patients, personals of non-busy units have been transferred in busier ones.

All these measures lead to major daily-life change sets that could be stressful. In the general population, it has been well documented that quarantine or confinement or isolation could lead to the occurrence of Post-Traumatic Stress Disorder (PTSD) syndrome in about 30% overall population. Importantly, high depressive symptoms have been reported in 9% of hospital staff. Numerous symptoms have been reported after quarantine or isolation such as emotional disturbance, depression, stress, low mood, irritability, insomnia, and post-traumatic stress symptoms.

In hospital setting, few studies have been performed for assessing the psychological impact of quarantine and isolation. However, two studies reported a high prevalence of burn-out syndrome (BOS) in ICU physician and PTSD syndrome and depression in ICU nurses. As the consequences of all the measures decided and applied during Covid-19 pandemic could be important on caregivers, the present study primarily aims at assessing the prevalence of PTSD syndrome in a large population of caregivers implied or not in Intensive Care Units. The secondary objective were 1) to assess the prevalence of severe depression and anxiety and BOS 2) to isolate potential factors associated with PTSD, severe depression, anxiety or BOS.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers (doctors senior and junior, nurses, aid nurses) involved in the staff (permanent or transient, full or partial time) of ICU patients during Covid-19 outbreak
* Approved to participate

Exclusion Criteria:

* Participation refusal
* No internet connection for responding to the questionnaire with REDCAP file

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers (doctors senior and junior, nurses, aid nurses) involved in the staff (permanent or transient, full or partial time) of ICU patients during Covid-19 outbreak
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder | 3-6 month after the Covid-19 outbreak
  PCL - 5 (Post-Traumatic Stress Disorder Checklist Scale, version DSM-5)

SECONDARY OUTCOMES:
anxiety and depression | 3-6 month after the Covid-19 outbreak
  HADS scale (Hospital Anxiety and Depression Scale)
Burn out | 3-6 month after the Covid-19 outbreak
  Score MBI (Burn out syndrome)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves LEFRANT, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (51):
- France (51):
  - Intensive Care Unit, CHU d'Amiens, Amiens
  - Intensive Care Unit, CHU d'Angers, Angers
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Hôpital Pellegrin, Bordeaux
  - Intensive care Unit CHU de Brest Hôpital Cavale Blanche, Brest
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - AP-HP, Hôpital Henri Mondor, Créteil
  - CHU de dijon, Dijon
  - CHU de Grenoble, Hôpital Michalon, La Tronche
  - AP_HP, Hôpital du Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Intensive Care Unit, CHRU de Lille, Lille
  - Intensive Care Unit, CHU de Limoges, Limoges
  - Hôpitaux civils de Lyon, Hôpital de la Croix Rousse, Lyon
  - Hôpitaux civils de Lyon, Hôpital Louis Pradel, Lyon
  - Hôpitaux civils de Lyon, Hôpital Edouard Herriot, Lyon
  - AP-HM, Hôpital Nord, Marseille
  - AP-HM, Hôpital Timone adultes, Intensive Care Unit, Marseille
  - AP-HM, Hôpital Timone adultes, Neurotraumatology, Marseille
  - AP-HM, Hôpital e la Conception, Marseille
  - CHU de Montpellier, Hôpital Guy de chauliac, Montpellier
  - CHU de Montpellier, Hôpital Lapeyronie, Montpellier
  - CHU de Montpellier, Hôpital St Eloi SAR B, Montpellier
  - CHU De Montpellier, Hôpital St Eloi-DAR B, Montpellier
  - CHU De Montpellier, Hôpital St Eloi, Montpellier
  - Intensive Care Unit, CHU de Mulhouse, Mulhouse
  - Intensive CAre Unit CHRU de Nancy, Hôpital Central, Nancy
  - Intensive Care Unit, CHU de Nantes, Hôtel Dieu, Nantes
  - Intensive Care Unit, CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Intensive care Unit CHU Nîmes, Nîmes
  - AP-HP, Hôpital de la Pitié, Paris
  - AP-HP, Hôpital Bichât, Paris
  - AP-HP, Hôpital Lariboisière, Paris
  - AP6HP, Hôpital St Loui, Paris
  - AP_HP, Hôpital G Pompidou, Paris
  - AP-HP, Hôpital St Antoine, Paris
  - CH de Perpignan, Perpignan
  - CHU de Bordeaux, Hôpital Haut Leveque, Pessac
  - Intensive care Unit, Hôpitaux civils de Lyon, Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Intensive care Unit CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de St Etienne, Hôpital Nord, Saint-Etienne
  - Intensive Care Unit, CHU de Nantes, Hôpital Laennec, Saint-Herblain
  - Intesive Care Unit CHRU de Strasbourg, Hôpital civil, Strasbourg
  - Intesive Care Unit CHRU de Strasbourg, Hôpital Hautepierre, Strasbourg
  - CHU de Toulouse, Toulouse
  - Intensive care unit CHU de Tours, Tours
  - Intensive CAre Unit CHRU de Nancy, Hôpital de Brabois, Vandœuvre-lès-Nancy
  - CH de Vesoul, Vesoul

REFERENCES:
- [Result] Roger C, Ling L, Petrier M, Elotmani L, Atchade E, Allaouchiche B, Aubrun F, Constantin JM, Dahyot-Fizelier C, Delhaye N, Dupont H, Fischer MO, Garnier M, Gayat E, Ichai C, Jaber S, Morel J, Plaud B, Rimmele T, Robin S, Saba R, Joynt GM, Lefrant JY, Fabbro-Peray P, Lipman J, Conejero I, Laupland K. Occurrences of post-traumatic stress disorder, anxiety, depression, and burnout syndrome in ICU staff workers after two-year of the COVID-19 pandemic: the international PSY-CO in ICU study. Ann Gen Psychiatry. 2024 Jan 3;23(1):3. doi: 10.1186/s12991-023-00488-5. PMID 38172994